CLINICAL TRIAL: NCT07073846
Title: Efficacy of Lidocaine-Dexmedetomidine Combination Therapy in Reducing Post-Operative Pain, Inflammatory Response, and Oxidative Stress in Patients Undergoing Bariatric Surgery
Brief Title: Effect of Lidocaine-Dexmedetomidine on Pain, Inflammation, and Oxidative Stress After Bariatric Surgery.
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Dulce Maria Rascon Martinez, Clinical Research Physician, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R-2025-3601-197
Record Dates: First submitted 2025-06-30; First posted 2025-07-18 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Morbid Obesity Requiring Bariatric Surgery; Postoperative Pain; Postoperative Pain Management; Postoperative Analgesia; Postoperative Adjuvant Treatment; Postoperative Inflammatory Markers; Postoperative Inflammatory Response
Keywords: Bariatric Surgery; Laparoscopic Sleeve Gastrectomy; Laparoscopic Gastric Bypass; Pain Management; Lidocaine-Dexmedetomidine; Multimodal Analgesia; Inflammatory Cytokines; Oxidative Stress; Opioid-sparing Anesthesia; Enhanced Recovery (ERAS); Postoperarive Oxidative Stress
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Lidocaine; Dexmedetomidine; Fluocinonide; Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomized, quadruple-masked, four-arm parallel design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomisation codes are generated in 13 permuted blocks of eight by an independent investigator who is not involved in patient care or outcome assessment. The codes are printed, placed in sequentially numbered, opaque, sealed envelopes, and handed to the study nursing team. Immediately before anaesthetic induction, a research nurse opens the next envelope and communicates the allocation to a second nurse-preparer (also independent from clinical care). This nurse draws up a visually identical 50 mL syringe containing lidocaine, dexmedetomidine, the fixed-dose combination (LIDEX), or 0.9 % saline, according to the code. Each syringe is labelled only with the participant ID and infusion rate. Emergency unblinding is allowed solely for patient-safety reasons and must be reported immediately to the Data and Safety Monitoring Board.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Lidocaine Infusion (LID) (Active Comparator): Intra-operative IV lidocaine 1 % at ≈ 1.5 mg·kg-¹·h-¹ (0.3 mL·kg-¹·h-¹). Infusion starts after induction and stops at skin closure; no post-operative infusion.
  Interventions: Drug: Intravenous Lidocaine infusion + Standard Anesthesia
- Dexmedetomidine Infusion (DEX) (Active Comparator): Intra-operative IV dexmedetomidine ≈ 0.3 µg·kg-¹·h-¹ (0.3 mL·kg-¹·h-¹) without loading dose, from induction to skin closure.
  Interventions: Drug: Intravenous Dexmedetomidine infusion + Standard Anesthesia
- Lidocaine + Dexmedetomidine (LIDEX) (Experimental): Concurrent IV lidocaine 1 % (1.5 mg·kg-¹·h-¹) plus dexmedetomidine (0.3 µg·kg-¹·h-¹) in the same syringe, administered from induction to skin closure.
  Interventions: Drug: Lidocaine + Dexmedetomidine Combination (LIDEX) + Standard Anesthesia
- Saline Placebo (Placebo Comparator): IV 0.9 % saline at 0.3 mL·kg-¹·h-¹ for the same duration as active arms; syringe identical in appearance.
  Interventions: Drug: 0.9 % Saline Placebo + Standard Anesthesia

INTERVENTIONS:
Drug: Intravenous Lidocaine infusion + Standard Anesthesia — Continuous IV infusion of lidocaine 1 % (10 mg mL-¹) at 0.3 mL kg-¹ h-¹ (≈ 1.5 mg kg-¹ h-¹) from induction of anaesthesia to skin closure. No loading bolus, no post-operative infusion.
  Other Names: Xylocaine®; Lignocaine
  Arms: Lidocaine Infusion (LID)
Drug: Intravenous Dexmedetomidine infusion + Standard Anesthesia — Continuous IV infusion of dexmedetomidine 1 µg mL-¹ at 0.3 mL kg-¹ h-¹ (≈ 0.3 µg kg-¹ h-¹) without loading dose, started after induction and stopped at skin closure. No post-operative infusion.
  Other Names: Precedex®; Dexdor®; DEX
  Arms: Dexmedetomidine Infusion (DEX)
Drug: Lidocaine + Dexmedetomidine Combination (LIDEX) + Standard Anesthesia — Single syringe containing lidocaine 1 % (10 mg mL-¹) + dexmedetomidine 1 µg mL-¹, infused IV at 0.3 mL kg-¹ h-¹ (delivering ≈ 1.5 mg kg-¹ h-¹ lidocaine + 0.3 µg kg-¹ h-¹ dexmedetomidine) from induction to skin closure.
  Other Names: LIDEX; Lidocaine-Dexmedetomidine cocktail; LID + DEX
  Arms: Lidocaine + Dexmedetomidine (LIDEX)
Drug: 0.9 % Saline Placebo + Standard Anesthesia — Volume-matched IV infusion of 0.9 % normal saline at 0.3 mL kg-¹ h-¹ for the same duration and through the same delivery line as active arms; identical syringe appearance.
  Other Names: Normal Saline; Sodium Chloride 0.9 %; Serum Saline; 0.9 % NaCl; Isotonic saline; Physiologic saline; Saline solution (IV)
  Arms: Saline Placebo

SUMMARY:
The goal of this randomized clinical trial is to find out whether giving an intravenous lidocaine + dexmedetomidine combination (LIDEX) during laparoscopic bariatric surgery can lower post-operative pain, inflammation, and oxidative stress in adults with obesity.

The main questions it aims to answer are:

* Pain control: Does LIDEX reduce pain 24 hours after surgery, as measured with the International Pain Outcomes Questionnaire (IPOQ)?
* Biomarkers: Does LIDEX lower blood levels of key inflammatory cytokines-interleukin-1 beta (IL-1β), interleukin-6 (IL-6), tumor necrosis factor-alpha (TNF-α), and interleukin-10 (IL-10)-and oxidative-stress markers-malondialdehyde (MDA), the reduced/oxidized glutathione ratio (GSH/GSSG), superoxide dismutase (SOD), and catalase-compared with the individual drugs or saline placebo?

Researchers will compare four groups: lidocaine alone, dexmedetomidine alone, LIDEX, and placebo (saline solution, a look-alike substance that contains no drug) to learn which approach works best.

Participants will:

* Receive an intravenous infusion of their assigned study drug(s) during surgery.
* Provide three small blood samples (before surgery, immediately after, and three hours after).
* Complete a short pain questionnaire (IPOQ) 24 hours after surgery.

DETAILED DESCRIPTION:
Obesity is associated with chronic low-grade inflammation and persistent oxidative stress. Laparoscopic bariatric surgery-although highly effective for weight reduction-triggers an acute inflammatory cascade and a burst of reactive oxygen species that can amplify post-operative pain and delay functional recovery.

Intravenous lidocaine stabilises voltage-gated Na+ channels, limits ectopic neuronal firing and inhibits neutrophil priming; it also down-regulates the release of pro-inflammatory cytokines in abdominal procedures. Dexmedetomidine, a highly selective α2-adrenergic agonist, produces sedation and analgesia while attenuating sympathetic outflow, thereby reducing surgical catecholamine surges and cytokine release. Pre-clinical and clinical synergy studies indicate that combining these two agents (LIDEX) can provide additive anti-hyperalgesic, anti-inflammatory and antioxidant effects without increasing cardiovascular risk when each is dosed within its established therapeutic window.

In this protocol, a weight-adjusted intra-operative infusion of lidocaine plus dexmedetomidine is administered during bariatric surgery and compared with each single agent and saline. Peri-operative venous samples are collected for mechanistic profiling of systemic inflammatory and redox responses, and patient-reported pain is captured after surgery using a validated instrument. Haemodynamic parameters are continuously monitored to detect potential lidocaine toxicity or dexmedetomidine-related bradycardia and hypotension; predefined rescue algorithms are applied if thresholds are exceeded.

The study is designed to clarify whether the LIDEX combination can blunt the acute inflammatory-oxidative surge thought to drive sustained pain and metabolic stress after bariatric surgery, thereby informing future enhanced-recovery protocols that integrate multimodal analgesia with metabolic optimisation strategies.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 - 60 years
* Male or female
* Elective laparoscopic bariatric surgery
* Post-operative pathway: post-anaesthesia care unit (PACU) followed by standard ward, with an expected in-hospital stay ≥ 24 h
* ASA physical-status II or III

Exclusion Criteria:

* Use of any loco-regional anaesthetic technique during the peri-operative period (transversus abdominis plane, paravertebral, spinal, epidural, erector spinae, or other abdominal wall blocks).
* Current substance abuse or illicit drug use.
* Previous abdominal surgery within the last 6 months.
* Known hypersensitivity or allergy to lidocaine, dexmedetomidine, amide local anaesthetics, or α₂-adrenergic agonists.
* Congestive heart failure, significant bradyarrhythmia, second- or third-degree atrio-ventricular block without pacemaker, severe hypotension, or current therapy with Class I/III anti-arrhythmic drugs.
* Estimated glomerular filtration rate (eGFR) < 60 mL min-¹ 1.73 m-² (moderate-to-severe renal impairment).
* Severe hepatic impairment (Child-Pugh C).
* Pregnancy or lactation.
* Chronic opioid consumption > 30 mg oral morphine equivalents per day for > 4 weeks
* Active seizure disorder, myasthenia gravis, or other neurologic disease contraindicating lidocaine infusion.
* Patient cannot communicate
* Patient does not want to fill in the questionnaire
* Participation in another interventional study within the past 30 days.
* Intra-operative conversion to open surgery.
* Insufficient biological sample for biomarker analysis.
* Premature discontinuation of the study drug during surgery for any reason that, in the judgement of the treating anaesthesiologist or investigators, prevents adequate exposure or assessment of safety variables (e.g., major haemorrhage > 200 mL, anaphylactic shock, failed intubation, inability to extubate, severe metabolic/respiratory acidosis, transfer to ICU while intubated).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of postoperative pain patient perception using the Spanish International Pain Outcomes Questionnaire (IPOQ). This questionnaire includes multiple items assessed on a numerical rating scale (NRS) from 0 to 10. | 24 hours post-operative
  * For most items (e.g., pain intensity, interference with activities, emotional impact), **higher scores indicate worse outcomes**.
  * For items such as pain relief and satisfaction, **higher scores indicate better outcomes**.
  Items include:
  * Highest and lowest pain intensity experienced since surgery
  * Proportion of time spent in pain
  * How pain limited physical activities (e.g., coughing, moving, walking)
  * Impact of pain on mood and emotional well-being
  * Adverse effects attributed to pain medication (e.g., nausea, dizziness)
  * Overall degree of pain relief obtained
  * Desire for additional analgesic treatment
  * Clarity and usefulness of information received about pain therapy
  * Extent of patient involvement in treatment decisions
  * Global satisfaction with pain management
  * Use of non-pharmacological methods for pain relief
  * Presence of pre-existing pain before hospital admission

SECONDARY OUTCOMES:
Change in pro-inflammatory cytokine (IL-1β, IL-6, TNF-α) and anti -inflammatory IL-10 panel | Day 0 - after anesthesia induction, end of surgery, and 3 hours postoperatively
  Serum concentrations of interleukin-1 beta (IL-1β), interleukin-6 (IL-6), and tumour necrosis factor-alpha (TNF-α) measured by multiplex ELISA (pg mL-¹). The primary comparison is the change from baseline and the area-under-curve (AUC₀-₃ h) across the four treatment arms; lower values indicate a reduced systemic inflammatory response.
Change in oxidative-stress marker panel (MDA, GSH/GSSG ratio, SOD, catalase, neutrophil respiratory burst) | Day 0 - after anesthesia induction, end of surgery, and 3 hours postoperatively
  Plasma malondialdehyde (MDA, µmol L-¹; TBARS assay), glutathione redox ratio (GSH/GSSG), superoxide-dismutase activity (SOD, U mL-¹) and catalase activity (U mL-¹) will be quantified with spectrophotometric/enzymatic methods. Neutrophil respiratory burst (reactive oxygen-species production) will be assessed by flow cytometry using DCFH-DA and expressed as mean fluorescence intensity (MFI). Change from baseline and the area-under-the-curve (AUC₀-3 h) will be compared across the four study arms; lower MDA/MFI and higher antioxidant indices indicate less oxidative stress.

CONTACTS AND LOCATIONS:
Overall Officials: Dulce María Rascón Martínez, Prof MD, MSc, Principal Investigator — Instituto Mexicano del Seguro Social; Arnulfo Calixto Flores, Prof MD, PhD, Principal Investigator — Instituto Mexicano del Seguro Social
Locations (2):
- Mexico (2):
  - Hospital de Especialidades Centro Medico Nacional Siglo XXI, Mexico City, Mexico City
  - Unidad Médica de Alta Especialidad Hospital de Especialidades del Centro Médico Nacional Siglo XXI, Mexico City, Mexico City

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that support the results reported in this study will be shared. This includes primary outcome data (IPOPQ responses), inflammatory cytokine levels (IL-1β, IL-6, TNF-α, IL-10), oxidative stress markers (MDA, SOD, catalase, GSH/GSSG ratio), and neutrophil respiratory burst results. All data will be anonymized and coded to protect participant confidentiality.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD will be available beginning 6 months after publication of the main study results in a peer-reviewed journal, and will remain available for up to 5 years after publication.
Access Criteria: The de-identified individual participant data (IPD) that support the results of this study will be available to any interested researchers.
  The data will be publicly accessible through an open-access Zenodo repository following publication of the main study results. No request or approval will be necessary. All data will be anonymized and will not contain any information that could identify participants. Supporting documents such as the protocol, statistical analysis plan, and informed consent form will also be available in the same repository.
URL: https://zenodo.org

REFERENCES:
- [Result] Xie D, Wang F, Wen W, Li H. Postoperative analgesic effect of intravenous coinjection of lidocaine and dexmedetomidine in gynaecological surgery: a systematic review and meta-analysis. BMJ Open. 2024 Dec 11;14(12):e091904. doi: 10.1136/bmjopen-2024-091904. PMID 39663167
- [Result] Rekatsina M, Theodosopoulou P, Staikou C. Effects of Intravenous Dexmedetomidine Versus Lidocaine on Postoperative Pain, Analgesic Consumption and Functional Recovery After Abdominal Gynecological Surgery: A Randomized Placebo-controlled Double Blind Study. Pain Physician. 2021 Nov;24(7):E997-E1006. PMID 34704710
- [Result] Zhang Y, Zhou Y, Hu T, Tong X, He Y, Li X, Huang L, Fu Q. Dexmedetomidine reduces postoperative pain and speeds recovery after bariatric surgery: a meta-analysis of randomized controlled trials. Surg Obes Relat Dis. 2022 Jun;18(6):846-853. doi: 10.1016/j.soard.2022.03.002. Epub 2022 Mar 9. PMID 35422388
- [Result] de Oliveira CMB, Coelho LMG, Valadao JA, Moura ECR, da Silva AAM, de Lima RC, Brunialti MKC, Salomao R, da Cunha Leal P, Sakata RK. Assessment of the Effect of Perioperative Venous Lidocaine on the Intensity of Pain and IL-6 Concentration After Laparoscopic Gastroplasty. Obes Surg. 2020 Oct;30(10):3912-3918. doi: 10.1007/s11695-020-04748-1. Epub 2020 Jun 12. PMID 32533519
- [Result] Xu S, Hu S, Ju X, Li Y, Li Q, Wang S. Effects of intravenous lidocaine, dexmedetomidine, and their combination on IL-1, IL-6 and TNF-alpha in patients undergoing laparoscopic hysterectomy: a prospective, randomized controlled trial. BMC Anesthesiol. 2021 Jan 6;21(1):3. doi: 10.1186/s12871-020-01219-z. PMID 33407156
- [Result] Lai Y, Chen Q, Xiang C, Li G, Wei K. Comparison of the Effects of Dexmedetomidine and Lidocaine on Stress Response and Postoperative Delirium of Older Patients Undergoing Thoracoscopic Surgery: A Randomized Controlled Trial. Clin Interv Aging. 2023 Aug 3;18:1275-1283. doi: 10.2147/CIA.S419835. eCollection 2023. PMID 37554513
- [Result] Chen X, Chen Q, Qin Z, Alam A, Zhao H, West R, Liu X, Li J, Li X, Yi B, Ma D, Gu J. Dexmedetomidine Attenuates Inflammation in Elderly Patients Following Major Hepatobiliary and Pancreatic Surgery: A Randomized Clinical Trial. Clin Interv Aging. 2024 May 29;19:981-991. doi: 10.2147/CIA.S455987. eCollection 2024. PMID 38827237
- [Result] Ohta Y, Miyamoto K, Kawazoe Y, Yamamura H, Morimoto T. Effect of dexmedetomidine on inflammation in patients with sepsis requiring mechanical ventilation: a sub-analysis of a multicenter randomized clinical trial. Crit Care. 2020 Aug 10;24(1):493. doi: 10.1186/s13054-020-03207-8. PMID 32778146
- [Result] Zhang J, Wang Z, Wang Y, Zhou G, Li H. The effect of dexmedetomidine on inflammatory response of septic rats. BMC Anesthesiol. 2015 May 1;15:68. doi: 10.1186/s12871-015-0042-8. PMID 25929655
- [Result] Avci O, Taskiran AS, Gundogdu O. Dexmedetomidina, un agonista de α2, incrementa el efecto analgésico de la morfina y reduce el desarrollo de tolerancia a la morfina suprimiendo el estrés oxidativo y la vía de señalización de TNF/IL-1 en ratas. Rev Esp Anestesiol Reanim
- [Result] Ge DJ, Qi B, Tang G, Li JY. Intraoperative Dexmedetomidine Promotes Postoperative Analgesia and Recovery in Patients after Abdominal Hysterectomy: a Double-Blind, Randomized Clinical Trial. Sci Rep. 2016 Feb 23;6:21514. doi: 10.1038/srep21514. PMID 26903197
- [Result] Kaye AD, Chernobylsky DJ, Thakur P, Siddaiah H, Kaye RJ, Eng LK, Harbell MW, Lajaunie J, Cornett EM. Dexmedetomidine in Enhanced Recovery After Surgery (ERAS) Protocols for Postoperative Pain. Curr Pain Headache Rep. 2020 Apr 2;24(5):21. doi: 10.1007/s11916-020-00853-z. PMID 32240402
- [Result] Lai YC, Wang WT, Hung KC, Chen JY, Wu JY, Chang YJ, Lin CM, Chen IW. Impact of intravenous dexmedetomidine on postoperative gastrointestinal function recovery: an updated meta-analysis. Int J Surg. 2024 Mar 1;110(3):1744-1754. doi: 10.1097/JS9.0000000000000988. PMID 38085848
- [Result] Jessen Lundorf L, Korvenius Nedergaard H, Moller AM. Perioperative dexmedetomidine for acute pain after abdominal surgery in adults. Cochrane Database Syst Rev. 2016 Feb 18;2(2):CD010358. doi: 10.1002/14651858.CD010358.pub2. PMID 26889627
- [Result] Lin S, Jin P, Shao C, Lu W, Xiang Q, Jiang Z, Zhang Y, Bian J. Lidocaine attenuates lipopolysaccharide-induced inflammatory responses and protects against endotoxemia in mice by suppressing HIF1alpha-induced glycolysis. Int Immunopharmacol. 2020 Mar;80:106150. doi: 10.1016/j.intimp.2019.106150. Epub 2020 Jan 17. PMID 31958741
- [Result] Lee JM, Suh JK, Jeong JS, Cho SY, Kim DW. Antioxidant effect of lidocaine and procaine on reactive oxygen species-induced endothelial dysfunction in the rabbit abdominal aorta. Korean J Anesthesiol. 2010 Aug;59(2):104-10. doi: 10.4097/kjae.2010.59.2.104. Epub 2010 Aug 20. PMID 20740215
- [Result] Gunaydin B, Demiryurek AT. Interaction of lidocaine with reactive oxygen and nitrogen species. Eur J Anaesthesiol. 2001 Dec;18(12):816-22. doi: 10.1046/j.1365-2346.2001.00931.x. PMID 11737181
- [Result] Castro I, Carvalho P, Vale N, Monjardino T, Mourao J. Systemic Anti-Inflammatory Effects of Intravenous Lidocaine in Surgical Patients: A Systematic Review and Meta-Analysis. J Clin Med. 2023 May 31;12(11):3772. doi: 10.3390/jcm12113772. PMID 37297968
- [Result] Beaussier M, Delbos A, Maurice-Szamburski A, Ecoffey C, Mercadal L. Perioperative Use of Intravenous Lidocaine. Drugs. 2018 Aug;78(12):1229-1246. doi: 10.1007/s40265-018-0955-x. PMID 30117019
- [Result] MacGregor RR, Thorner RE, Wright DM. Lidocaine inhibits granulocyte adherence and prevents granulocyte delivery to inflammatory sites. Blood. 1980 Aug;56(2):203-9. No abstract available. PMID 7397378
- [Result] Paterson HM, Cotton S, Norrie J, Nimmo S, Foo I, Balfour A, Speake D, MacLennan G, Stoddart A, Innes K, Cameron S, Aucott L, McCormack K. The ALLEGRO trial: a placebo controlled randomised trial of intravenous lidocaine in accelerating gastrointestinal recovery after colorectal surgery. Trials. 2022 Jan 28;23(1):84. doi: 10.1186/s13063-022-06021-5. PMID 35090535
- [Result] Ahn E, Kang H, Choi GJ, Park YH, Yang SY, Kim BG, Choi SW. Intravenous lidocaine for effective pain relief after a laparoscopic colectomy: a prospective, randomized, double-blind, placebo-controlled study. Int Surg. 2015 Mar;100(3):394-401. doi: 10.9738/INTSURG-D-14-00225.1. PMID 25785316
- [Result] Eipe N, Gupta S, Penning J. Intravenous lidocaine for acute pain: an evidence-based clinical update. BJA Educ. 2016 Sep 1;16(9):292-8.
- [Result] Baysal Z, Togrul T, Aksoy N, Cengiz M, Celik H, Boleken ME, Kaya M, Yavuz G. Evaluation of total oxidative and antioxidative status in pediatric patients undergoing laparoscopic surgery. J Pediatr Surg. 2009 Jul;44(7):1367-70. doi: 10.1016/j.jpedsurg.2008.11.031. PMID 19573663
- [Result] Tsuchiya M, Sato EF, Inoue M, Asada A. Open abdominal surgery increases intraoperative oxidative stress: can it be prevented? Anesth Analg. 2008 Dec;107(6):1946-52. doi: 10.1213/ane.0b013e318187c96b. PMID 19020142
- [Result] Mieszczanski P, Gorniewski G, Ziemianski P, Cylke R, Lisik W, Trzebicki J. Comparison between multimodal and intraoperative opioid free anesthesia for laparoscopic sleeve gastrectomy: a prospective, randomized study. Sci Rep. 2023 Aug 4;13(1):12677. doi: 10.1038/s41598-023-39856-2. PMID 37542100
- [Result] Ivascu R, Torsin LI, Hostiuc L, Nitipir C, Corneci D, Dutu M. The Surgical Stress Response and Anesthesia: A Narrative Review. J Clin Med. 2024 May 20;13(10):3017. doi: 10.3390/jcm13103017. PMID 38792558
- [Result] Torensma B, Hany M, Bakker MJS, van Velzen M, In 't Veld BA, Dahan A, Swank DJ. Correction to: Cross-Sectional E-survey on the Incidence of Pre- and Postoperative Chronic Pain in Bariatric Surgery. Obes Surg. 2023 Jan;33(1):211. doi: 10.1007/s11695-022-06395-0. No abstract available. PMID 36463344
- [Result] Iamaroon A, Tangwiwat S, Nivatpumin P, Lertwacha T, Rungmongkolsab P, Pangthipampai P. Risk Factors for Moderate to Severe Pain during the First 24 Hours after Laparoscopic Bariatric Surgery While Receiving Intravenous Patient-Controlled Analgesia. Anesthesiol Res Pract. 2019 Oct 3;2019:6593736. doi: 10.1155/2019/6593736. eCollection 2019. PMID 31687018
- [Result] Garduno-Lopez AL, Acosta Nava VM, Castro Garces L, Rascon-Martinez DM, Cuellar-Guzman LF, Flores-Villanueva ME, Villegas-Sotelo E, Carrillo-Torres O, Vilchis-Samano H, Calderon-Vidal M, Islas-Lagunas G, Richard Chapman C, Komann M, Meissner W, Baumbach P, Zaslansky R. Towards Better Perioperative Pain Management in Mexico: A Study in a Network of Hospitals Using Quality Improvement Methods from PAIN OUT. J Pain Res. 2021 Feb 15;14:415-430. doi: 10.2147/JPR.S282850. eCollection 2021. PMID 33623424
- [Result] De Oliveira GS Jr, Duncan K, Fitzgerald P, Nader A, Gould RW, McCarthy RJ. Systemic lidocaine to improve quality of recovery after laparoscopic bariatric surgery: a randomized double-blinded placebo-controlled trial. Obes Surg. 2014 Feb;24(2):212-8. doi: 10.1007/s11695-013-1077-x. PMID 24036842
- [Result] Tufanogullari B, White PF, Peixoto MP, Kianpour D, Lacour T, Griffin J, Skrivanek G, Macaluso A, Shah M, Provost DA. Dexmedetomidine infusion during laparoscopic bariatric surgery: the effect on recovery outcome variables. Anesth Analg. 2008 Jun;106(6):1741-8. doi: 10.1213/ane.0b013e318172c47c. PMID 18499604